CLINICAL TRIAL: NCT01096901
Title: Weight Loss to Reduce Breast Cancer Risk Factors
Brief Title: Choose to Lose for Women-Weight Loss to Reduce Breast Cancer Risk Factors
Acronym: CTL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Suzanne Phelan, Principal Investigator, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CP-CTL; CP-EFI
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive behavioral weight loss (Active Comparator): The group will be implemented to induce a 6% weight loss over 3 months. The lessons will follow protocols from the Look AHEAD trial and Diabetes Prevention Program. This behavioral program has been shown to promote long-term weight loss and a reduction in diabetes and cardiovascular risk factors, and is based on the social cognitive theory.
  Interventions: Behavioral: Behavioral Weight loss
- Education and Support Control group (No Intervention): Participants in this group will receive support and education about healthy eating and activity with lessons based on the Look AHEAD support and education control condition. Participants will attend monthly closed group meetings and meetings will be designed to promote retention but not weight loss.

INTERVENTIONS:
Behavioral: Behavioral Weight loss — Intervention groups will meet weekly for 12 weeks. Weekly meetings will focus on weight loss in women age 30-45 through behavioral weight loss topics. These topics are designed with the Look AHEAD protocols.
  Arms: Comprehensive behavioral weight loss

SUMMARY:
This study is investigating the changes in specific hormone levels in women age 30-45 after a 12 week weight loss intervention.

DETAILED DESCRIPTION:
In sum, excess body weight and inactivity have emerged as strong avoidable causes of postmenopausal breast cancer, with the greatest potential for primary prevention occurring during the premenopausal years. However, surprisingly, no study to date has examined the effects of a standard behavioral weight loss intervention on breast cancer risk markers in premenopausal women. Understanding the effects of weight loss in premenopausal women is a critical next step in existing research and will inform the development of future breast cancer primary prevention programs. The purpose of this study is to determine the feasibility of recruiting, treating, and retaining 20 overweight/obese women in a 12-week randomized control trial examining feasibility and effects of a behavioral weight loss program on breast cancer risk markers in premenopausal women. Participants will be randomly assigned to either a 12-week comprehensive behavioral weight loss program (n=10) or control condition (n=10). All women will be assessed at baseline and after 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* Age 30-45
* Current BMI of >25
* English or Spanish speaking
* 5th grade reading level
* Menstrual regularity, defined as menstrual cycle length of 27-31 and < 1 missed period within the past 12 months.

Exclusion Criteria:

* Current use or recent (< 6 months) use of oral contraceptives, hormones, or other hormone-influencing medications
* Pregnant, lactating or planning pregnancy in the next 12 weeks
* Unwilling and able to location for intervention visits.
* Serious medical condition requiring the supervision of a physician for exercise and diet
* History of eating disorder
* History of or current use of drugs
* Current treatment for serious psychological disorder
* Donation of blood within past 6 weeks.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Weight loss for one group | 3 months
  One group in this randomized study will be focused on weight loss during a 3 month period. The goal is to acheive a 6% weight loss during this time. Specific blood draws will be conducted pre and post weight loss to measure any hormonal changes due to this weight loss.

SECONDARY OUTCOMES:
Increased physical activity | 3 months
  The secondary objective in this study is to increase participant activity level to help reduce the risks of certain cancers. As well as increase the overall health of these participants.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Phelan, PhD., Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States